CLINICAL TRIAL: NCT00378924
Title: Cardiology Biobank Registry
Status: Recruiting | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Other Study IDs: IRB00000343; 950-2003 (Other: Other)
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 60 cc of blood will be obtained from the participant. Blood will be processed and stored in -80F freezers as plasma, serum, extracted DNA and whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In the present study, investigators intend to establish a large database of cardiovascular patients. More specifically, investigators will create a database of approximately 12,000 cardiac catheterization and heart failure patients from Emory University Hospital, the Emory Clinic, Emory University Hospital Midtown, Grady Memorial Hospital, Atlanta VA Medical Center, Organized/Planned Community Events in the Atlanta Metropolitan area, held at places of Worship, local Community Centers, shopping Malls, doctor's Offices and Health Clinics and any other miscellaneous locations, e.g. Parks, Leisure centers, Conference centers.

Once the data has been collected, investigators will run a variety of statistical analyses to which will help us to learn more about the factors that cause various cardiovascular diseases such as coronary heart disease, angina, heart failure, hypertension, and stroke. The statistical analyses will also help us to understand how these diseases can be treated more effectively.

By collecting a large amount of data on a large number of cardiovascular patients, investigators will be able to analyze, with a great deal of precision, those factors that influence the onset, course, and treatment of cardiovascular disease. The results of these precise analyses can then be used to help optimize clinical efforts to prevent and treat cardiovascular disease.

DETAILED DESCRIPTION:
Over the last several decades, scientists have made great progress in their understanding of cardiovascular disease. Nevertheless, much remains to be learned about the causes, course, and treatment of cardiovascular disease. In order to learn more about this topic, it is important to establish large databases of cardiovascular patients. These databases allows scientists to investigate, in a rigorous and precise manner, those factors that influence cardiovascular disease.

In the present study, investigators intend to establish a large database of cardiovascular patients. More specifically, investigators will create a database of approximately 12,000 cardiac catheterization and heart failure patients from Emory University Hospital, the Emory Clinic, Emory University Hospital Midtown, Grady Memorial Hospital, Atlanta VA Medical Center, Organized/Planned Community Events in the Atlanta Metropolitan area, held at places of Worship, local Community Centers, shopping Malls, doctor's Offices and Health Clinics and any other miscellaneous locations, e.g. Parks, Leisure centers, Conference centers.

Investigators will collect a large amount of data on these patients. Data to be collected will include information on:

Medical record data, including imaging Patient questionnaire data DNA and other biochemical data obtained and/or generated from patient blood samples or cheek (buccal) swabs Non-invasive measurements of blood pressure, heart rate and studies relating to assessment of the health of arteries

The data noted above will be collected by:

administering questionnaires/interviews to the patients accessing the medical records of the patients collecting blood samples from patients which will be analyzed by laboratories for their biochemical content.

Once the data has been collected, investigators will run a variety of statistical analyses to which will help us to learn more about the factors that cause various cardiovascular diseases such as coronary heart disease, angina, heart failure, hypertension, and stroke. The statistical analyses will also help investigators to understand how these diseases can be treated more effectively.

How the Research Will Advance Scientific Knowledge/Human Health:

By collecting a large amount of data on a large number of cardiovascular patients, investigators will be able to analyze, with a great deal of precision, those factors that influence the onset, course, and treatment of cardiovascular disease. The results of these precise analyses can then be used to help optimize clinical efforts to prevent and treat cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

1. All hospital and clinic patients aged 18 years and older
2. Patients with active cardiovascular disease including but not limited to

   1. Ischemic Heart Disease
   2. Heart Failure and Cardiomyopathies
   3. Peripheral Vascular Disease
   4. Valve disease
   5. Adult Congenital Heart disease
   6. Electrophysiological Disorders
3. Any Atlanta metropolitan area resident aged 18 and above in satisfactory physical health and able to tolerate a blood draw or buccal swab.

Exclusion Criteria:

1. Significant Documented Anemia (Hemoglobin <8 g/dL)
2. Blood transfusions within past 3 weeks
3. Active Cancer (non-skin cancers)
4. Enrollment against doctor recommendation
5. Patient not able to provide consent including but not limited to:

   1. Intubated and critically unwell patients
   2. Dementia
   3. Alzheimer's disease
   4. Moderate to severe alcohol or drug abuse
   5. Against religious beliefs (e.g. Jehovah's witness

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population & patients presenting to the hospital
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2003-12; Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
All cause death | Continuous

SECONDARY OUTCOMES:
Cardiovascular death | Continuous
Re-hospitalization for heart failure | Continuous

OTHER OUTCOMES:
Myocardial Infarction | Continuous
Stroke | Continuous

CONTACTS AND LOCATIONS:
Overall Officials: Arshed A Quyyumi, MD, Principal Investigator — Emory School Of Medicine
Locations (1):
- Emory School Of Medicine, Atlanta, Georgia, United States